CLINICAL TRIAL: NCT00604695
Title: A Randomized Trial Evaluating Low-Dose IntraCoronary AdjunctivE Tenecteplase During Primary PCI for ST-Elevation Myocardial Infarction (ICE T)
Brief Title: A Safety/Efficacy Study of Intra-coronary Tenecteplase During Balloon Angioplasty to Treat Heart Attacks
Acronym: ICE T-TIMI 49
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C. Michael Gibson, MS, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, C. Michael Gibson, MS, MD, Sponsor-Investigator, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N3770S
Record Dates: First submitted 2008-01-07; First posted 2008-01-30 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-08

CONDITIONS: Acute Myocardial Infarction
Keywords: ST-Elevation Myocardial Infarction; Acute Myocardial Infarction; No Reflow
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tenecteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Two (4mg) doses of tenecteplase
  Interventions: Drug: Tenecteplase
- 2 (Placebo Comparator): Two (4mL) doses of sterile saline
  Interventions: Drug: Sterile Saline

INTERVENTIONS:
Drug: Tenecteplase — Intracoronary injection of IV tenecteplase.
  Arms: 1
Drug: Sterile Saline — Intracoronary injection of IV sterile saline
  Arms: 2

SUMMARY:
The primary objective of this study is to gather preliminary data regarding the angiographic efficacy of the administration of low-dose adjunctive intracoronary (IC) tenecteplase during balloon angioplasty for heart attacks.

We hypothesize that low-dose IC tenecteplase will enhance the breakdown of blood clots at the site of the culprit lesion leading to reduced damage to the heart muscle.

DETAILED DESCRIPTION:
The primary objective of this study is to gather preliminary data regarding the angiographic efficacy of the administration of low-dose adjunctive intracoronary (IC) tenecteplase during primary percutaneous coronary intervention (PCI) for ST-segment elevation myocardial infarction (STEMI). Efficacy will be assessed by measurements of both the angiographic characteristics of the culprit lesion as well as by measurements of epicardial flow and myocardial perfusion in the territory of the infarct-related artery. This study will also evaluate the safety of administering low-dose IC tenecteplase to subjects undergoing primary PCI for STEMI treated with standard therapy (aspirin, clopidogrel, and glycoprotein IIb/IIIa inhibitors). Safety endpoints include the incidence of death, recurrent myocardial infarction (MI), abrupt vessel closure, subacute stent thrombosis, and TIMI major and minor bleeding events.

Prompt reperfusion therapy with primary PCI in patients with STEMI improves clinical outcomes through salvage of myocardial tissue. The proposed pilot trial is a randomized, placebo-controlled trial to evaluate the effectiveness and safety of adjunctive low-dose IC tenecteplase in conjunction with standard medical therapy during primary PCI for STEMI. We hypothesized that low-dose IC tenecteplase will enhance fibrinolysis at the site of the culprit lesion leading to reduced microvascular dysfunction. As reduced dose tenecteplase will be injected directly into the coronary artery increasing local concentration of the drug with minor systemic effects, an improved safety profile is also expected from this mode of administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (men or women) at least 18 years and less than 75 years of age and
* Ischemic discomfort ≥20 minutes and ≤6 hours of duration and
* ST elevation ≥1mm (≥0.1mV) in two contiguous limb leads OR ≥2mm (≥0.2mV) in two contiguous precordial leads and
* Occluded infarct-related artery (TIMI Flow Grade 0 or 1) at the time of coronary angiography and
* Planned primary PCI within 2 hours of hospital presentation and
* Planned or concomitant use of aspirin, clopidogrel, unfractionated heparin, and Glycoprotein IIb/IIIa inhibition with intent to stent the infarct-related artery and
* Informed consent able to be obtained

Exclusion Criteria:

CLINICAL

* Age ≥75 years
* Maximal systolic blood pressure <80 mmHg AFTER initial fluid and/or pressor resuscitation.
* Uncontrolled hypertension (SBP >180 OR DBP >110) at time of enrollment.
* Cardiac arrest or arrhythmia requiring chest compressions or cardiopulmonary resuscitation.
* Known pregnancy.

BIOCHEMICAL

* Known thrombocytopenia (platelet count <100,000)
* Known severe renal insufficiency (creatinine >4.0 mg/dL).

INCREASED BLEEDING RISK

* Active internal bleeding
* Recent (<3 months) gastrointestinal hemorrhage
* Recent intracranial or intraspinal surgery, trauma, major surgery, or biopsy of a parenchymal organ (< 1 month)
* Known coagulopathy, platelet disorder, or history of thrombocytopenia
* Current warfarin therapy
* Known neoplasm
* Any known history of transient ischemic attack, cerebrovascular accident, or active intracranial pathology including arteriovenous malformation or aneurysm

MEDICATIONS

* Administration of a fibrinolytic agent within 72 hours
* Known allergy or contraindication to fibrinolytics OR aspirin OR heparin OR clopidogrel

ANGIOGRAPHIC

* Left Main Coronary artery culprit lesion
* Ostial culprit lesion (ostium of LAD, LCX, or RCA).
* Lesion in non-native coronary artery (e.g. saphenous vein graft, arterial conduit graft)
* Subjects requiring urgent coronary artery bypass grafting

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Michael Gibson, MS, MD, Principal Investigator — Brigham and Women's Hospital
Locations (8):
- United States (8):
  - Northeast Georgia Heart Center, PC, Gainesville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory University, Decatur, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Crittenton Hospital Medical Center, Rochester, Michigan
  - Heart Consultants, PC, Freemont, Nebraska
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Gibson CM, Kumar V, Gopalakrishnan L, Singh P, Guo J, Kazziha S, Devireddy C, Pinto D, Marshall JJ, Stouffer GA, Mavromatis K, Grip L, Bainey KR; TIMI & PERFUSE Study Group. Feasibility and Safety of Low-Dose Intra-Coronary Tenecteplase During Primary Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction (ICE T-TIMI 49). Am J Cardiol. 2020 Feb 15;125(4):485-490. doi: 10.1016/j.amjcard.2019.11.018. Epub 2019 Nov 20. PMID 31870492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study randomized 40 primary percutaneous coronary intervention (PPCI) patients from 6 hospitals in the United States. The patients were given either a volume matched bolus of intracoronary (IC) tenecteplase (TNK) (4 mg; n=20) or IC saline placebo (4 mg; n=16) before and following PPCI. 4 subjects were randomized but did not receive 1st bolus.
Groups:
- Active Treatment: Two (4mg) doses of tenecteplase
- Placebo Control: Two (4mL) doses of sterile saline
Period: Overall Study
Arm/Group | Active Treatment | Placebo Control
Started | 20 | 20
Completed | 20 | 16
Not Completed | 0 | 4
Not completed — Did not receive first bolus. | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (7.6) | 55.6 (8.9) | 55.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent Diameter Stenosis of the Culprit Lesion Following the First Bolus of Study Drug Prior to Primary Percutaneous Coronary Intervention
Time Frame: Following the First Bolus of Study Drug Prior to Primary Percutaneous Coronary Intervention
Population: Of the 20 patients randomized to the treatment arm, 4 patients did not meet the inclusion criteria of Thrombolysis In Myocardial Infarction (TIMI) Flow Grade(TFG) 0/1.
  Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo) and 3 patients did not meet the inclusion criteria of TFG 0/1.
Measure: Median (Inter-Quartile Range); unit: Percent diameter stenosis
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 16 | 13
Percent diameter stenosis | 100 [83 to 100] | 100 [100 to 100]

2. Secondary Outcome: Number of Patients With Decrease in Thrombus Grade in the Culprit Artery Following the First Bolus of Study Drug Prior to Primary Percutaneous Coronary Intervention
Time Frame: Following the First Bolus of Study Drug Prior to Primary Percutaneous Coronary Intervention
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 16 | 13
participants | 7 | 2

3. Secondary Outcome: Number of Patients With Thrombolysis In Myocardial Infarction (TIMI) Myocardial Perfusion Grade (TMPG) of 2 or 3 in the Territory of the Culprit Artery Following Primary Percutaneous Coronary Intervention Prior to Second Bolus of the Study Drug
Description: Thrombolysis In Myocardial Infarction (TIMI) Myocardial Perfusion Grade (TMPG) of 2 or 3 in the territory of the culprit artery
Time Frame: Following Primary Percutaneous Coronary Intervention Prior to Second Bolus of the Study Drug
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 16 | 13
participants | 8 | 8

4. Secondary Outcome: Measurements of Flow Velocity in the Culprit Artery in Terms of Corrected Thrombolysis In Myocardial Infarction (TIMI) Frame Count (cTFC)
Description: Corrected Thrombolysis In Myocardial Infarction (TIMI) Frame Count (cTFC) in the culprit artery
Time Frame: Following Primary Percutaneous Coronary Intervention Prior to Second Bolus of the Study Drug
Population: Of the 20 patients in treatment arm, 4 did not meet the inclusion criteria of TIMI Flow Grade(TFG) 0/1 and cTFC could not be obtained in 4 patients Of the 20 patients in placebo arm, 4 did not receive the first bolus (drug or placebo) and 3 patients did not meet the inclusion criteria of TFG 0/1. cTFC could not be obtained in 3 patients
Measure: Median (Inter-Quartile Range); unit: Corrected TIMI Frame Count (cTFC)
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 12 | 10
Corrected TIMI Frame Count (cTFC) | 26 [21 to 33] | 14 [10 to 24]

5. Secondary Outcome: Number of Patients With Hyperemic Flow in the Culprit Artery. That is Corrected Thrombolysis In Myocardial Infarction (TIMI) Frame Count (cTFC) of Less Than 14
Description: Corrected Thrombolysis In Myocardial Infarction (TIMI) Frame Count (cTFC) of less than 14
Time Frame: Following Primary Percutaneous Coronary Intervention Prior to Second Bolus of the Study Drug
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 12 | 10
participants | 1 | 5

6. Secondary Outcome: Safety Endpoint: Number of Patients Who Developed Thrombolysis In Myocardial Infarction (TIMI) Minor Bleeding
Time Frame: Through 30days following PPCI
Population: Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo)
Measure: Number; unit: participants
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 20 | 16
participants | 1 | 0

7. Secondary Outcome: Safety Endpoint: Number of Patients Who Developed Thrombolysis In Myocardial Infarction (TIMI) Minimal Bleeding
Time Frame: Through 30days following primary percutaneous coronary intervention
Population: Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo)
Measure: Number; unit: participants
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 20 | 16
participants | 4 | 2

8. Secondary Outcome: Safety Endpoint: Number of Patients Who Developed Cardiac Arrhythmias
Time Frame: Through 30days following primary percutaneous coronary intervention
Population: Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo)
Measure: Number; unit: participants
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 20 | 16
participants | 1 | 2

9. Secondary Outcome: Safety Endpoint: Number of Deaths
Time Frame: Through 30days following primary percutaneous coronary intervention
Population: Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo)
Measure: Number; unit: participants
Arm/Group | Active Treatment | Placebo Control
Number analyzed (Participants) | 20 | 16
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 30-days following primary percutaneous coronary intervention
Description: Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Arm/Group | Active Treatment | Placebo Control
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/16
Other Adverse Events (participants affected / at risk) | 14/20 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=20) | Placebo Control (N=16)
Erosive Gastritis (Gastrointestinal disorders) | 1 | 0 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Dressler's syndrome (Cardiac disorders) | 0 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Death (General disorders) | 1 | 0 — Cause of death unknown. Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=20) | Placebo Control (N=16)
Anemia (Blood and lymphatic system disorders) | 1 | 0 — Pre-existing anemia. Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Ventricular Tachycardia (Cardiac disorders) | 1 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Pancreatitis (Gastrointestinal disorders) | 1 | 0 — Pre-existing chronic pancreatitis. Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Clostridium difficile infection (Infections and infestations) | 1 | 0 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Right hand and finger numbness (Injury, poisoning and procedural complications) | 0 | 1 — Primary percutaneous coronary intervention was performed via radial approach. Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Right groin cellulitis (Injury, poisoning and procedural complications) | 0 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Urinary tract infection (Infections and infestations) | 1 | 0 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Pre-existing asthma. Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Allergic reaction to Bactrim (Immune system disorders) | 0 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Allergic reaction to Lisinopril (Immune system disorders) | 0 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Bleeding (Injury, poisoning and procedural complications) | 5 | 2 — Bleeding at the site of insertion of catheter. Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Hypotension (Cardiac disorders) | 1 | 0 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Chest pain (Cardiac disorders) | 1 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
Back pain (General disorders) | 0 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).
High grade Atrio-Ventricular Block (Cardiac disorders) | 1 | 1 — Of the 20 patients randomized to the placebo arm, 4 patients did not receive the first bolus (drug or placebo).

LIMITATIONS AND CAVEATS:
This pilot study was not adequately powered to exclude a modest increase in bleeding events. Study drug could not be administered to 4 patients and 7 patients were excluded for not meeting the inclusion criteria of TIMI Flow Grade 0/1 at enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator shall furnish Sponsor with copy of any proposed publication for review/comment prior to submission for publication, at least thirty (30) days prior to submission for manuscripts and at least fifteen (15) days prior to submission for abstracts. Institution agrees to delete information identified by Sponsor as Confidential Information prior to submission for publication.